CLINICAL TRIAL: NCT07297316
Title: Comparison of Immediate Therapeutic Effects of 3% Diquafosol and 2% Rebamipide in Dry Eye Disease
Brief Title: Immediate Therapeutic Effects of Diquafosol and Rebamipide in Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Kukje Pharma (Other)
Responsible Party: Principal Investigator, Dong Hyun Kim, Principal Investigator, Korea University Anam Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2022AN0535
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — diquafosol; rebamipide

STUDY DESIGN:
Intervention Model Description: This is a paired-eye design study, where patients received 3% diquafosol in one eye and 2% rebamipide in the contralateral eye.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R) DQS, L) REB (Other): This is a paired-eye design study. Patients were randomly assigned to receive 3% diquafosol in the right eye and 2% rebamipide in the contralateral left eye, with the treatment assignment blinded to the examiner and patients.
  Interventions: Drug: 3% diquafosol (right eye) and 2% rebamipide (left eye)
- R) REB, L) DQS (Other): This is a paired-eye design study. Patients were randomly assigned to receive 3% diquafosol in the left eye and 2% rebamipide in the contralateral right eye, with the treatment assignment blinded to the examiner and patients.
  Interventions: Drug: 2% rebamipide (right eye) and 3% diquafosol (left eye)

INTERVENTIONS:
Drug: 3% diquafosol (right eye) and 2% rebamipide (left eye) — 3% diquafosol was instilled in the right eye and 2% rebamipide in the left eye.
  Arms: R) DQS, L) REB
Drug: 2% rebamipide (right eye) and 3% diquafosol (left eye) — 2% rebamipide was instilled in the right eye and 3% diquafosol in the left eye.
  Arms: R) REB, L) DQS

SUMMARY:
This study compares the immediate therapeutic and mucin-secreting effects 30 minutes after instillation of 3% diquafosol and 2% rebamipide in dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* patients 19 years or older
* complaint of at least one dry eye symmptom and tear breakup time < 7 seconds

Exclusion Criteria:

* Sjogren's syndrome
* prescription history of systemic steroids or immunosuppressants
* prior ocular surgery within six months of enrollment
* treatment with diquafosol or rebamipide eye drops within 2 weeks of enrollment
* treatment with punctal plug within 1 month of enrollment
* intraocular pressure exceeding 25mmHg
* usage of contact lens during the study
* active ocular infection
* pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) score | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  Unit: points
tear breakup time (TBUT) | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  Unit: Seconds
ocular staining score (OSS) | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  National Eye Institute Scale, 0-15
tear meniscus height (TMH) | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  Unit: mm
lipid layer thickenss (LLT) | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  Unit: nm
corneal sensitivity (esthesiometer) | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  Unit: mm

SECONDARY OUTCOMES:
tear MUC1 concentration | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  measured using enzyme-linked immunosorbent assay (ELISA)
tear MUC5AC concentration | Before instillation of eyedrops, and 30 minutes after instillation of eyedrops
  measured using enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not openly available due to reasons of sensitivity and may available from the corresponding author upon reasonable request.